CLINICAL TRIAL: NCT02631785
Title: Fear Conditioning, Extinction and Its Recall in Anxious Youth: Identifying Neuro- Cognitive Abnormalities and Their Relation to Pediatric Anxiety Treatment Outcomes
Brief Title: Fear Conditioning, Extinction and Its Recall in Anxious Youth
Acronym: FCPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Haifa (Other)
Collaborators: HaEmek Medical Center, Israel (Other); Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Tomer Shechner, Principal Investigator, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 97-15; 1377/14 (Other Grant/Funding Number: Israel Science Foundation); 618534 (Other Grant/Funding Number: CIG-2013)
Record Dates: First submitted 2015-12-02; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric Anxiety Disorders
Keywords: ANXIETY; CBT; fMRI; Fear conditioning; Fear extinction
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anxious group (Experimental): Youth diagnosed with anxiety disorder will receive Cognitive Behavioral Therapy for reducing anxiety symptoms.
  Interventions: Other: Cognitive Behavioral Therapy
- Control group (No Intervention): Healthy youth will be recruited for comparison but their participant in the study will not include intervention.

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — Psychologists will deliver the "COPING CAT" treatment for reducing anxiety symptoms. It is a manualized treatment that was extensively used before. The treatment will include 10- 14 sessions, mostly individual but also two parents meetings. All the treatments will occur in the Department of Psychology in Haifa University as a part of a clinical trial. The treatment will take place in a room that was designed for this purpose fully equipped with cameras, microphone and double sided mirror. All sessions will be audio and video recorded and will be closely monitored by the PI. To increase protocol adherence and verify the adequacy of the treatment delivered, all clinicians will complete routine forms with the content of each session.
  Other Names: CBT
  Arms: Anxious group

SUMMARY:
The proposed research aims to isolate brain-based information-processing mechanisms implicated in perturbed fear learning and extinction characteristic of pediatric anxiety.

The study will focus on the therapeutic relevance of dysfunction in fear learning and extinction for treatment by examining the associations between brain functioning and response to exposure intervention in anxious children.

DETAILED DESCRIPTION:
Anxiety disorders are the most common form of pediatric psychopathology, affecting 5 - 20% of children and adolescents. Despite therapeutic advances, treatment-resistance remains high, and progress towards early detection of at-risk populations and more effective treatments has stalled. Although some anxiety disorders are transient, recent studies suggest that pediatric anxiety disorders commonly persist into adulthood. Because anxiety disorders are costly and debilitating conditions that are very often associated with other severe psychopathology such as substance abuse, depression and suicidality, there is an imperative need to identify risk and resilience factors that moderate pediatric anxiety and improve treatment.

Fear conditioning and resistance to extinction are two domains that have been implicated in the etiology and maintenance of anxiety disorders. Indeed, one of the most effective treatment for pediatric and adult anxiety disorders, exposure therapy, relies profoundly on extinction learning. The proposed research plan will investigate the neural correlates of aberrant fear conditioning and extinction processes in children and adolescents with anxiety disorders.

The proposed research aims to isolate brain-based information-processing mechanisms implicated in perturbed fear learning and extinction characteristic of pediatric anxiety. A fMRI study using a novel age-appropriate fear conditioning-extinction paradigm are proposed. The study will delineate perturbed psychological and psychophysiological response to fear conditioning and isolate neuro-cognitive mechanisms mediating extinction recall in anxious and non-anxious children. Three weeks after completing fear conditioning and extinction task in the psychophysiology lab, participants will return to complete an fMRI extinction-recall task quantifying responses to extinguished CS blends. Two major hypotheses will be examined: a) anxious children will exhibit perturbations during extinction as measured by psychophysiology indexes and self-reported fear compared to non-anxious children; b) less activation in ventromedial prefrontal cortex (vmPFC) is expected in anxious, relative to healthy, children during extinction-recall. Furthermore, the study will focus on the therapeutic relevance of dysfunction in fear learning and extinction for treatment by examining the associations between vmPFC function and response to exposure intervention in anxious children. Lower levels of vmPFC activation prior to exposure therapy and larger pre-to-post-treatment changes in vmPFC activity are expected to be associated with better response to exposure therapy.

ELIGIBILITY:
Research Group:

Inclusion Criteria:

* diagnosis of Separation Anxiety Disorder, Social Phobia or Generalized Anxiety Disorder.

Exclusion Criteria:

* other psychiatry diagnose (not include depression and ADHD)
* currently in psychological treatment
* psychiatry medication

Control group:

Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

* any psychiatry diagnose.
* currently in psychological treatment
* psychiatry medication

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
fMRI Bold signal | 2 years
  analysis of brain activation

SECONDARY OUTCOMES:
Autonomous measures- skin conductance response (SCR) | 2 years
  skin conductance response (SCR) will be recorded from the participant's hand using two standard electrodes attached to the participants' palm.
Self report of anxiety | 2 years
  participants will rate their level of fear during watching stimuli
Autonomous measures-Fear-Potentiated Startle | 2 years
  will be measured through electromyography (EMG) of the eye-blink reflex following a puff of air to the forehead.
Anxiety symptom- SCARED | 2 years
  • The Screen for Child Anxiety Related Emotional Disorders (SCARED) - the SCARED is a self-report measure that assesses different types of anxiety based on criteria in the DSM-IV. Specifically, the SCARED was developed as a screening tool for generalized anxiety disorder, separation anxiety disorder, panic disorder, social phobia, and school phobia. The SCARED has been reported to have robust reliability and validly (Birmaher et al., 1997).
Anxiety symptoms- ADIS | 2 years
  The Anxiety Disorder Interview Schedule (ADIS) - is a well validated semi-structured diagnostic interview, suitable for measuring all anxiety disorders as listed in the DSM-IV as well as mood disorders and attention deficit hyperactivity disorder, in children from 7-17 years of age (Silverman & Albano, 1996). The interview has two versions, one for children (ADIS-C) and one for parents (ADIS-P), and both have good inter-rater and high test-retest reliability (Silverman, Saavedra, & Pina, 2001). In standard ADIS procedures, a child receive a diagnosis when a specified amount of criteria are met the child or parent reports substantial interference (4 or higher on a scale from 0 to 8). The combined diagnosis represents a sum of the diagnoses of the child and the parent interview
Anxiety symptoms- CGI | 2 years
  Clinical Global Impression scale (CGI). The CGI scale requires clinicians to rate the overall severity of their patient's illness at the time of assessment relative to the clinician's experience with patients having the same diagnosis. This scale yields three different measures: severity of illness, global improvement, and the efficacy index. The ratings range from 1 (very much improved) to 7 (very much worse) (Busner & Targum, 2007).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - University of Haifa, Haifa
  - Weizmann Institue of Science, Rehovot

REFERENCES:
- [Background] Beesdo K, Knappe S, Pine DS. Anxiety and anxiety disorders in children and adolescents: developmental issues and implications for DSM-V. Psychiatr Clin North Am. 2009 Sep;32(3):483-524. doi: 10.1016/j.psc.2009.06.002. PMID 19716988
- [Background] Shechner T, Hong M, Britton JC, Pine DS, Fox NA. Fear conditioning and extinction across development: evidence from human studies and animal models. Biol Psychol. 2014 Jul;100:1-12. doi: 10.1016/j.biopsycho.2014.04.001. Epub 2014 Apr 16. PMID 24746848
- [Background] Shechner T, Britton JC, Ronkin EG, Jarcho JM, Mash JA, Michalska KJ, Leibenluft E, Pine DS. Fear conditioning and extinction in anxious and nonanxious youth and adults: examining a novel developmentally appropriate fear-conditioning task. Depress Anxiety. 2015 Apr;32(4):277-88. doi: 10.1002/da.22318. Epub 2014 Nov 27. PMID 25427438
- [Background] Walkup JT, Albano AM, Piacentini J, Birmaher B, Compton SN, Sherrill JT, Ginsburg GS, Rynn MA, McCracken J, Waslick B, Iyengar S, March JS, Kendall PC. Cognitive behavioral therapy, sertraline, or a combination in childhood anxiety. N Engl J Med. 2008 Dec 25;359(26):2753-66. doi: 10.1056/NEJMoa0804633. Epub 2008 Oct 30. PMID 18974308
- [Result] Britton JC, Grillon C, Lissek S, Norcross MA, Szuhany KL, Chen G, Ernst M, Nelson EE, Leibenluft E, Shechner T, Pine DS. Response to learned threat: An FMRI study in adolescent and adult anxiety. Am J Psychiatry. 2013 Oct;170(10):1195-204. doi: 10.1176/appi.ajp.2013.12050651. PMID 23929092